CLINICAL TRIAL: NCT03447496
Title: Multi-center Study on Surgical Treatment for the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children
Brief Title: Surgical Treatment for the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children
Acronym: JCHLCF
Status: Completed | Type: Observational
Sponsor: Shunyou Chen (Other)
Responsible Party: Sponsor-Investigator, Shunyou Chen, Director,Head of Orthopaedics, The Fuzhou No 2 Hospital
Organization: The Fuzhou No 2 Hospital (Other)
Other Study IDs: Shunyou Chen
Record Dates: First submitted 2018-01-31; First posted 2018-02-27 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-02

CONDITIONS: Lateral Condyle Fractures,Humerus,JakobⅡ Classification,Reduction
MeSH Terms: interventions — Closed Fracture Reduction; Open Fracture Reduction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Closed reduction: The children were treated with closed reduction.
  Interventions: Procedure: Closed reduction
- Open reduction: The children were treated with open reduction.
  Interventions: Procedure: Open reduction

INTERVENTIONS:
Procedure: Closed reduction — The children were treated with closed reduction.
  Groups: Closed reduction
Procedure: Open reduction — The children were treated with Open reduction.
  Groups: Open reduction

SUMMARY:
Multi-center Study on Surgical Treatment for the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children.

DETAILED DESCRIPTION:
The Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children that were treated with closed or open reduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fractures that met these criteria, underwent definitive surgery and had complete clinical and radiographic follow up until fracture union at either institution were included in this study.

Exclusion Criteria:

* Pathologic fractures, and fractures in patients with osteogenesis imperfecta, neuromuscular disorders or any systemic disease that was associated with a predisposition to fractures or altered fracture healing were excluded.

Max Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Surgical Treatment for the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Radiographic union | Up to 12 weeks.
  Radiographic union in surgical treatment for the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children.

SECONDARY OUTCOMES:
Fracture displacement | Up to 12 weeks.
  Fracture displacement in surgical treatment for the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children.

OTHER OUTCOMES:
Functional clinical scores | Through study completion, an average of 1 year.
  Dhillon scoring system for the outcome of the Displaced JakobⅡ Classification Humerus Lateral Condylar Fractures in Children.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Shunyou, Phd, Study Director — The Fuzhou No 2 Hospital
Locations (1):
- Shunyou Chen, Fuzhou, Fujian, China